CLINICAL TRIAL: NCT01062321
Title: Role of Cytokines in Hepatitis E Virus Infection During Pregnancy
Status: Completed | Type: Observational
Sponsor: Maulana Azad Medical College (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Ashok Kumar, Director Professor, Maulana Azad Medical College
Other Study IDs: 5/7/239/07/RHN
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2011-07

CONDITIONS: Hepatitis; Cytokines; Pregnancy
Keywords: Hepatitis E Virus; Cytokines; Pregnancy
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis-E, Pregnant & Non-pregnant: Pregnant,Acute Viral Hepatitis, Fulminant Hepatic Failure

SUMMARY:
Hepatitis E virus is a public health problem in several countries of the world where safe drinking water is a problem. HEV is an exclusive cause of epidemic hepatitis in general population. HEV infection occurs most frequently in rainy season. The disease affects mainly young adults in the age of 15-40 years.HEV viral infection is of particular concern in pregnancy. It is a potential disaster for mother and child. HEV infection during pregnancy is fulminant and fatal especially if it occurs in third trimester. The mortality in the second trimester is around 20% and reaches upto 45% in the third trimester.

DETAILED DESCRIPTION:
The study will include pregnant women with acute viral hepatitis and fulminant hepatic failure (jaundice). The women with FHF will be recruited from the medical wards and antenatal wards as all such patients are routinely admitted in the hospital.

The pregnant women with acute viral hepatitis will be recruited either from antenatal clinic and medical outpatient, or from the medical and antenatal wards because pregnant women with AVH are admitted if they have serum bilirubin levels > 15- 20 mg / dl, persistently high bilirubin levels for more than 2-3 weeks, abnormal prothrombin time, evidence of progression of the disease, need parenteral therapy (because of excessive vomiting).

The enrolled subjects will be evaluated on the basis of a pre-designed and pre-tested proforma with respect to history and clinical examination, obstetrics examination and ultrasonography. Ten ml venous blood sample will be drawn from the patient at the time of enrollment detection of hepatotropic viruses (Various serological markers of hepatitis will be done which includes: IgM anti-HAV, HBsAg, IgM anti-HBc, HBeAg, anti-HCV Ab and IgM anti-HEV would be done using commercially available ELISA kits and Extraction of HEV-RNA from serum will be done) & levels of cytokines (IL-6, TGF-beta, IFN-g and TNF-α). All the subjects will be followed- up till delivery. The promoter region of cytokine gene will be amplified by PCR in appropriate reaction conditions using suitable sets of primers. PCR product will be used for studying the polymorphisms by restriction fragment length polymorphism.

The control group would comprise of age and POG matched healthy asymptomatic pregnant women

Follow up

All participants will be followed up till delivery for obstetrical complications, medical complications and pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria of acute viral hepatitis - Patients having acute self-limited disease and a serum aspartate aminotransferase elevation of at least 5 fold or clinical jaundice or both.
2. Diagnostic criteria of acute liver failure - When after a typical acute onset, the patient becomes deeply jaundiced and goes into hepatic encephalopathy within 4 weeks of the onset of disease with no past history of chronic liver disease.
3. Diagnostic criteria of Hepatitis E infection - The serum sample showing HEV IgM positivity and/or HEV-RNA positivity would be considered as HEV infected cases.

Exclusion Criteria:

1. Patients with co-infection with other hepatitis virus. 2. Patients with any other associated diseases. 3. Patients with history of pre-existing liver disease.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women of 18-40 years with jaundice and Healthy pregnant women as controls
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To correlate the levels of cytokines and its genes polymorphisms with the severity of hepatitis in HEV and non-HEV pregnant women. | 3 years

SECONDARY OUTCOMES:
To correlate the outcome of pregnancy with the levels of maternal cytokines and its genes polymorphisms. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ashok Kumar, MD, Principal Investigator — Maulana Azad Medical College, New Delhi-110002
Locations (1):
- Dr. Ashok Kumar, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Dahiya M, Kumar A, Kar P, Gupta RK, Kumar A. Acute viral hepatitis in third trimester of pregnancy. Indian J Gastroenterol. 2005 May-Jun;24(3):128-9. No abstract available. PMID 16041115
- [Result] Beniwal M, Kumar A, Kar P, Jilani N, Sharma JB. Prevalence and severity of acute viral hepatitis and fulminant hepatitis during pregnancy: a prospective study from north India. Indian J Med Microbiol. 2003 Jul-Sep;21(3):184-5. PMID 17643015
- [Result] Hussaini SH, Skidmore SJ, Richardson P, Sherratt LM, Cooper BT, O'Grady JG. Severe hepatitis E infection during pregnancy. J Viral Hepat. 1997 Jan;4(1):51-4. doi: 10.1046/j.1365-2893.1997.00123.x. PMID 9031065
- [Result] Navaneethan U, Al Mohajer M, Shata MT. Hepatitis E and pregnancy: understanding the pathogenesis. Liver Int. 2008 Nov;28(9):1190-9. doi: 10.1111/j.1478-3231.2008.01840.x. Epub 2008 Jul 25. PMID 18662274
- [Result] Barrett S, Collins M, Kenny C, Ryan E, Keane CO, Crowe J. Polymorphisms in tumour necrosis factor-alpha, transforming growth factor-beta, interleukin-10, interleukin-6, interferon-gamma, and outcome of hepatitis C virus infection. J Med Virol. 2003 Oct;71(2):212-8. doi: 10.1002/jmv.10472. PMID 12938195